CLINICAL TRIAL: NCT00245050
Title: A Double-Blind Randomized Trial of Pyridoxine Versus Placebo for the Prevention of Doxil-Related Palmar-Plantar Erythrodysesthesia (Hand-Foot Syndrome)
Brief Title: Pyridoxine in Preventing Hand-Foot Syndrome in Patients Who Are Receiving Liposomal Doxorubicin for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CASE5Y03; P30CA043703 (NIH); CASE5Y03 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer; Drug/Agent Toxicity by Tissue/Organ; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: drug/agent toxicity by tissue/organ; fallopian tube cancer; peritoneal cavity cancer; recurrent ovarian epithelial cancer; recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Breast Neoplasms, Male | interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyridoxine (Experimental): Arm I: Patients receive doxorubicin HCl liposome IV 40 mg/m2 over 1 hour on day 1 and oral pyridoxine 100 mg twice daily on days 1-28.
  Interventions: Dietary Supplement: pyridoxine hydrochloride; Drug: doxorubicin HCL liposome
- Placebo (Placebo Comparator): Arm II: Patients receive doxorubicin HCl liposome IV 40 mg/m2 over 1 hour on day 1 and oral placebo twice 100 mg daily on days 1-28.
  Interventions: Drug: Placebo; Drug: doxorubicin HCL liposome

INTERVENTIONS:
Dietary Supplement: pyridoxine hydrochloride — Arm I: Patients receive doxorubicin HCl liposome IV 40 mg/m2 over 1 hour on day 1 and oral pyridoxine twice 100 mg daily on days 1-28.
  Arms: Pyridoxine
Drug: Placebo — Arm II: Patients receive doxorubicin HCl liposome IV 40 mg/m2 over 1 hour on day 1 and oral placebo 100 mg twice daily on days 1-28.
  Arms: Placebo
Drug: doxorubicin HCL liposome — IV, 40mg/m2

SUMMARY:
RATIONALE: Pyridoxine (vitamin B6) may prevent or lessen hand-foot syndrome caused by chemotherapy. It is not yet known whether pyridoxine is more effective than a placebo in preventing hand-foot syndrome.

PURPOSE: This randomized clinical trial is studying pyridoxine to see how well it works compared to a placebo in preventing hand-foot syndrome in patients who are receiving liposomal doxorubicin for recurrent ovarian, fallopian tube, or peritoneal cancer, metastatic breast cancer, or advanced endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of pyridoxine vs placebo in preventing palmar-plantar erythrodysesthesia (PPE) in patients receiving doxorubicin HCl liposome for recurrent ovarian, fallopian tube, or peritoneal cavity cancer, metastatic breast cancer, or advanced endometrial cancer.
* Compare quality of life in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind study. Patients are stratified according to cancer type (ovarian, fallopian tube, or peritoneal cavity cancer vs breast cancer vs endometrial cancer). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxorubicin HCl liposome IV 40mg/m2 over 1 hour on day 1 and oral pyridoxine 100 mg twice daily on days 1-28.
* Arm II: Patients receive doxorubicin HCl liposome IV 40mg/m2 over 1 hour on day 1 and oral placebo 100 mg twice daily on days 1-28.

In both arms, treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients who develop grade 2-3 palmar-plantar erythrodysesthesia despite dose reduction of doxorubicin HCl liposome are unblinded and removed from the study (for patients in arm I) OR receive oral pyridoxine twice daily beginning day 1 of the next planned therapy (for patients in arm II).

Quality of life is assessed at baseline and after every third course of therapy.

After completion of study treatment, patients are followed periodically for 6 months.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Recurrent ovarian, fallopian tube, or peritoneal cavity cancer
  * Metastatic breast cancer
  * Advanced endometrial cancer
* Planning to receive chemotherapy with doxorubicin HCl liposome at a dose of 40 mg/m^2
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Not specified

Menopausal status:

* Not specified

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* AST and ALT ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* Bilirubin normal

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* Ejection fraction ≥ 50% by MUGA or 2-D echocardiogram
* No history of cardiac disease
* No New York Heart Association class II-IV heart disease
* No clinical evidence of congestive heart failure

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No active infection requiring antibiotics
* No history of hypersensitivity reaction attributed to a conventional formulation of doxorubicin HCl or doxorubicin HCl liposome and any of its components
* No other invasive malignancy within the past 5 years except nonmelanoma or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic or immunologic agents for this cancer

Chemotherapy

* Recovered from prior chemotherapy

  * Alopecia or neuropathy allowed
* No prior doxorubicin HCl liposome
* Other concurrent chemotherapy allowed provided palmar-plantar erythrodysesthesia is not one of the side effects of the therapy

  * No concurrent cytarabine, fluorouracil, liposomal daunorubicin, or capecitabine
  * No concurrent pre-medication with corticosteroids as part of the chemotherapy regimen

Endocrine therapy

* See Chemotherapy
* At least 3 weeks since prior and no concurrent oral or topical corticosteroids
* At least 1 week since prior hormonal therapy for this cancer

  * Concurrent hormone replacement therapy allowed

Radiotherapy

* At least 3 weeks since prior radiotherapy for this cancer and recovered

Surgery

* Recovered from prior surgery

Other

* At least 3 weeks since prior and no other concurrent forms of pyridoxine except what is included in a multivitamin
* No prior anticancer treatment that contraindicates study treatment
* No concurrent amifostine or other protective agents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-04; Primary Completion 2008-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian von Gruenigen, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (8):
- United States (8):
  - Geauga Regional Hospital, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the outpatient gynecologic oncology clinics at University Hospitals from May 2004 to December 2007.
Pre-assignment Details: Patients were required to have discontinued corticosteroid therapy at least three weeks prior to enrollment and no corticosteroids were allowed for the duration of the trial. Patients must have discontinued pyridoxine therapy at least three weeks prior to enrollment.
Groups:
- Pyridoxine: Arm I: Patients receive doxorubicin HCl liposome IV 40mg/m2 over 1 hour on day 1 and oral pyridoxine 100 mg twice daily on days 1-28.
- Placebo: Arm II: Patients receive doxorubicin HCl liposome IV 40mg/m2 over 1 hour on day 1 and oral placebo 100 mg twice daily on days 1-28.
Period: Overall Study
Arm/Group | Pyridoxine | Placebo
Started | 18 | 16
Completed | 15 | 14
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyridoxine | Placebo | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.4) | 65.9 (11.0) | 64.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Palmar-plantar Erythrodysesthesia (PPE)
Description: Patients were monitored weekly with phone calls from the research nurse and monthly at clinic visits for overall (including pyridoxine) and specific doxorubicin HCl liposome related toxicities using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
Time Frame: Treatment repeats every 4 weeks for up to 6 courses in the absence of unacceptable toxicity.
Population: Patients were evaluable for PPE/HFS(Hand-Foot Syndrome) incidence and toxicity assessment if they received at least one course of chemotherapy. Intention to treat analysis was used.
Measure: Number; unit: participants
Arm/Group | Pyridoxine | Placebo
Number analyzed (Participants) | 15 | 14
participants
  Grade 1 HFS | 2 | 3
  Grade 2 HFS | 3 | 3
  Grade 3 HFS | 3 | 1
Statistical Analysis 1: Comparison: Pyridoxine vs Placebo; Based on published literature, it is estimated that the incidence of HFS for all grades is 49%. A decrease of 50% or more in the incidence of HFS in patients receiving pyridoxine would be of clinical significance. A sample size of 27 patients per group was chosen as this would allow us to detect a difference between HFS incidence of 49% and 11.5% (alpha=0.05, two-sided, power=0.80). Interim analysis was conducted after 30 patients were enrolled and had evaluable HFS assessment data; Test type: Superiority or Other; p < 0.05, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.536 to 2.16]

2. Secondary Outcome: Quality of Life (QOL) as Measured by Functional Assessment of Cancer Therapy (FACT-G)
Description: QOL was measured with the FACT-G questionnaire following the third course of doxorubicin HCl liposome before the patient was seen by the treating physician and before chemotherapy was administered. The FACT-G, version 4, is a 27-item core questionnaire evaluating the domains of physical, functional, family-social, and emotional well-being (PWB, FWB, SWB, EWB). Total score ranges from 0-108 and higher scores indicate better QOL.
Time Frame: After Cycle 3 of chemotherapy (on average at 3 months)
Measure: Mean (Standard Deviation); unit: Total scores on FACT-G scale
Arm/Group | Pyridoxine | Placebo
Number analyzed (Participants) | 15 | 14
Total scores on FACT-G scale | 84.9 (10.2) | 84.4 (9.5)
Statistical Analysis 1: Comparison: Pyridoxine vs Placebo; Test type: Superiority or Other; p = 0.916, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Patients were monitored weekly with phone calls from the research nurse and monthly at clinic visits for overall (including pyridoxine) and specific PLD-related toxicities using the NCI CTCAE, version 3.0
Arm/Group | Pyridoxine | Placebo
Serious Adverse Events (participants affected / at risk) | 8/15 | 6/14
Other Adverse Events (participants affected / at risk) | 13/15 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyridoxine (N=15) | Placebo (N=14)
Allergy/immunologic (Immune system disorders) | 0 (0) | 1 (1)
Blood/bone marrow (Blood and lymphatic system disorders) | 1 (4) | 2 (4)
Constitutional symptoms (General disorders) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage/bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphatics (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Metabolic/laboratory (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neurology (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal/genitourinary (Renal and urinary disorders) | 0 (0) | 0 (0)
Vascular (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyridoxine (N=15) | Placebo (N=14)
Blood/bone marrow (Blood and lymphatic system disorders) | 7 (36) | 8 (42)
Constitutional symptoms (General disorders) | 7 (7) | 5 (8)
Gastrointestinal (Gastrointestinal disorders) | 9 (11) | 5 (7)
Hepatic/pancreas (Hepatobiliary disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 1 (3)
Lymphatics (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Metabolic/laboratory (Metabolism and nutrition disorders) | 1 (3) | 1 (6)
Musculoskeletal/soft tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neurology (Nervous system disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 5 (5) | 2 (6)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Renal/genitourinary (Renal and urinary disorders) | 2 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
Interim analysis was conducted after 30 patients were enrolled and had evaluable PPE assessment data. Due to decreased accrual and similar PPE rates between groups, the trial was closed for enrollment after the interim analyses was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No